CLINICAL TRIAL: NCT05605366
Title: Minocycline in Neurocognitive Outcomes - Sickle Cell Disease
Acronym: MINO-SCD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Kristine Karkoska, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-0375
Record Dates: First submitted 2022-10-20; First posted 2022-11-04 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-09

CONDITIONS: Sickle Cell Disease; Cognitive Impairment; Cognitive Decline; Cognitive Change; Cognitive Dysfunction; Cognitive Deficit; Neuroinflammatory Response
Keywords: sickle cell disease; benign hematology; cognitive dysfunction; neuroinflammation
MeSH Terms: conditions — Anemia, Sickle Cell; Cognitive Dysfunction; Cognition Disorders; Neuroinflammatory Diseases | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment arm (1) (Experimental): This arm will receive 200mg of minocycline in a single capsule per day.
  Interventions: Drug: Minocycline
- Treatment arm (2) (Active Comparator): This arm will receive 300 mg of minocycline in a single capsule per day. This capsule is identical in size and appearance as the 200 mg capsule
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): This arm will receive the placebo which is similar in size and appearance as the 200 mg and 300 mg capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — Minocycline is a second-generation tetracycline antibiotic with good central nervous system penetration and anti-neuroinflammatory effect.
  Arms: Treatment arm (1); Treatment arm (2)
Drug: Placebo — This is capsule that is identical in size and appearance as the drug, but without active drug ingredient.
  Arms: Placebo

SUMMARY:
Sickle cell disease (SCD) is a common, inherited blood disorder that primarily affects people of African Ancestry. It has a lot of complications including neurological complications. The neurological complications of SCD are particularly devastating and lead to cognitive decline even in the absence of overt brain injury. In such cases, it is thought that inflammation in the brain maybe partly responsible for the cognitive decline.

The main reasons for this research study are to see 1) how safe and 2) how well minocycline works to try to stop/reverse cognitive decline in people with SCD. People with SCD are at risk for changes in their brain over time that can cause problems with learning, memory, and attention. Part of the reason for this is inflammation within the brain. Minocycline may be able to stop these brain changes by stopping this brain inflammation.

Minocycline is a second-generation tetracycline antibiotic that has been shown to both inhibit neuroinflammation and improve cognitive function in a variety of neurodegenerative and psychiatric disorders but has not yet been studied in SCD. We are proposing here, a pilot double-blinded, randomized controlled trial to examine the tolerability and early efficacy of minocycline in adults with SCD at two dosing regimens (200 mg and 300 mg daily) versus placebo over one year. Participants will undergo a neuropsychological exam using the NIH Toolbox Cognition Battery at both study enrollment and exit (after one year) to assess for changes/stability of cognition. Participants will receive monthly phone calls/text messages to assess for adverse events and will be seen every three months for pill counts and routine laboratory monitoring. The primary outcome will be a comparison of adverse events across the two dosing strategies versus placebo. Early evidence for cognitive benefit will also be assessed from the results of the NIH Toolbox.

DETAILED DESCRIPTION:
Study Overview: This is a pilot study examining tolerability of low (200 mg daily) and high (300 mg daily) oral minocycline in adults with SCD compared to placebo. We will aim to enroll and randomize 30 adults with SCD and monitor for 12 months. Preliminary data regarding cognition will be obtained at baseline and 12 months, safety/laboratory monitoring will be incorporated into clinical care at 3 month intervals, with monthly phone calls and/or text messaging to inquire about any adverse event that may have occurred since the last clinic visit.

Inclusion/Exclusion: Adults (age ≥ 18 years old) with SCD (HbSS and HbS-β0thalassemia genotypes only) who are followed at the University of Cincinnati Medical Center's SCD clinic are eligible to participate. As hydroxyurea is the standard-of-care in SCD, individuals on hydroxyurea will be included. The exclusion criteria are as follows: 1) adults with other SCD genotypes (HbSC or HbS- β+thalassemia), 2) individuals with a history of overt stroke or other known neurological disorder, 3) premature birth before 30 weeks gestation, 4) monthly therapy with chronic blood transfusions, 5) coexisting autoimmune condition due to an elevated risk for autoimmune-related complications with tetracyclines, and 6) tetracycline allergy. Study members will approach eligible individuals at their regularly scheduled hematology visits to assess for interest and complete consent. All study-related procedures will be performed by the University of Cincinnati's specifications.

Dose Justification: The proposed dosing is based on previous double-blind placebo-controlled studies of minocycline use in neuropsychiatric disorders. In the Minocycline in Alzheimer Disease Efficacy (MADE) trial 200 mg daily resulted in no difference in adverse event or drug discontinuation rates compared to placebo, in contrast to 400 mg daily, which had significantly higher rates of dermatologic and gastrointestinal side effects.22 In patients with schizophrenia, minocycline 200 mg daily was associated with improvement in cognition at 3 months compared to placebo with no difference in adverse events.19, 38 A larger study of 204 patients with schizophrenia receiving minocycline 300 mg daily found no difference in adverse events between the minocycline and placebo groups.21 Finally, patients with clinical isolated syndrome (a precursor to multiple sclerosis) who received minocycline 200 mg daily saw a decrease in conversion to multiple sclerosis at six months; however, the rates of trial withdrawal and adverse events, including rash, dizziness, and dental discoloration, were higher in the minocycline versus placebo arm.39 Thus, it is unclear whether 200 mg daily or 300 mg daily is the optimal dose in adult SCD.

Cognitive Assessments: Participants will complete the NIH Toolbox: Cognition Battery, the Consortium to Establish a Registry for Alzheimer's disease Verbal Learning Test (CERAD-VLT), and the Complex Taylor Figure at baseline visit and 12-month follow up. The NIH Toolbox, a cognitive outcome measure designed for epidemiologic research and clinical trials, is administered via tablet application with automated scoring and was validated in a diverse cohort of 476 participants ages 3-85 years.40 The NIH Toolbox has previously been utilized in pediatric SCD participants, detecting the decreased inhibitory control, processing speed, and cognitive flexibility which have been observed in previous studies.41 To compliment the NIH Toolbox we will utilize the CERAD-VLT to assess verbal learning, including episodic memory.42 Lastly, children with SCD can have significant visual spatial dysfunction as the result of cerebral infarcts, we anticipate the same might be the case with the adults and as such, we will assess visual spatial ability using the Complex Taylor Figure tool.8, 43 Intervention, Measurements, & Data Collection: Upon enrollment, all participants will undergo neuropsychological assessment at baseline using the tools described above. All participants will also undergo a baseline symptom assessment, physical examination, peripheral oxygen saturation, and laboratory analysis, including complete blood count (CBC) with differential, reticulocyte count, complete metabolic panel (CMP), fetal hemoglobin (HbF), thyroid function tests, and spot urine microalbumin. If any laboratory analysis had been completed within two weeks prior to enrollment, this will not be repeated. Individuals will then be randomized to receive minocycline 200 mg daily, minocycline 300 mg daily, or placebo via a random number generator. Both the patient and investigator will be blinded to the enrollment status. Participants will return for pill counts, laboratory examination, and physical exam every three months. Participants will also fill out a standardized assessment regarding their health and any side effects monthly; this will be administered via RedCAP survey either through phone call/text message or via tablet application and can be completed at home during the months between study visits. The study visits will be timed ideally with routine clinical follow ups in the Hoxworth Clinic, but with all study-related procedures taking place in the Schubert Research Clinic at Cincinnati Children's Hospital Medical Center. Participants will also undergo the following labs every three months during study visits: CBC, CMP, reticulocyte count, and HbF; these will not be repeated if obtained clinically within two weeks of the study visit date. Thyroid function tests and urine microalbumin will be collected every six months. Study enrollees will be followed for a period of 12 months from their day of starting either the drug or placebo. Participants will then repeat the components of the baseline studies, including the neuropsychological assessment. Participants and study investigators will have the option to be unblinded to each participant's study arm.

Study Duration: The total study duration will be two years; we expect 6 months for patient recruitment/randomization followed by 12 months of therapy and another 6 months for data analysis/publication.

Statistical Analysis and Power Calculations: If the outcome distributions of the data are close to normal distributions, Student's t test (paired or unpaired) or chi-square test will be performed for descriptive statistics. If the outcome fails the normality tests, Mann-Whitney rank sum test will be used. Additionally, when comparing all 3 groups, ANOVA and/or non-parametric Kruskal-Wallis tests will be used when necessary. Post hoc testing on ANOVA will be done by multiple pairwise comparison procedures using the Holm-Sidak method. When repeated measurements of the outcomes are observed, mixed effect linear or generalized linear models will be used. Our sample size calculations indicate that with the proposed sample size (n=7 patients/group), we will be able to reach 80% power to detect an effect size of 1.6 between groups for continuous outcomes (Aim 2 - rate of decline in neurocognition); and an effect size of around 0.95 (using arcsine scale) for binary outcomes (Aim 1 - adverse events). If the true effect sizes are smaller, our study will not be powered to detect statistical significance between groups; however, the insights generated (especially for our primary outcome of tolerability) from this study will be useful for planning a larger phase II/III efficacy trial. All estimated differences in the outcomes, p-values and the corresponding 95% confidence intervals will be provided. P values below 0.05 will be reported as significant. All data will be analyzed using R, Version 3.3.3 (R Core Team 2012).

Rigor and Reproducibility: The NIH Toolbox: Cognition Battery is easily administered via tablet application and has been validated in a diverse racial, ethnic, and socioeconomic population; the scores are normalized to those of a standard neuropsychological battery (including full scale intelligence quotient) with a mean = 100 and standard deviation = 15. Thus, Toolbox results can be compared to those of participants of future studies.

Strengths, Limitations, & Alternative Approaches: This study is unique in that it is the first assessment of safety and early efficacy for the use or potential long-term use of minocycline in individuals with sickle cell disease to slow the expected rate of cognitive decline. This study is strengthened using two dosing strategies, both of which have proven efficacious and safe in other neurologic and psychiatric disorders. In addition, as this will be a pilot for a large phase II/III study, only those individuals with the HbSS and HbS- β0thalassemia genotypes will be included, which will be the expected population for the proposed larger trial and will limit confounding from differences in SCD genotypes. The primary limitation for this study is its small sample size; the study may not be powered to evaluate efficacy of minocycline to slow the expected rate of neurocognitive decline in SCD; however, the findings could be informative especially with regards to short and possibly long-term tolerability of minocycline. Another limitation is the potential for drop out and noncompliance with the study drug; however, we will attempt to minimize these risks with pairing study visits with routine clinical visits and with a monetary honorarium of $20 for the completion of study enrollment procedures, every three-month study visits, and the final 12 month study procedures. We will aim to recruit ten patients in each arm for a total of 30 patients to account for a 30% drop out rate. Finally, if recruitment becomes difficult, we will limit the minocycline arm to the 300 mg dosing strategy only.

ELIGIBILITY:
Inclusion Criteria:

Adults (age ≥ 18 years old) with SCD (HbSS and HbS-β0thalassemia genotypes only) who are followed at the University of Cincinnati Medical Center's SCD clinic are eligible to participate. As hydroxyurea is the standard-of-care in SCD, individuals on hydroxyurea will be included

Exclusion Criteria:

1. adults with other SCD genotypes (HbSC or HbS- β+thalassemia),
2. individuals with a history of overt stroke or other known neurological disorder,
3. premature birth before 30 weeks gestation,
4. monthly therapy with chronic blood transfusions,
5. coexisting autoimmune condition due to an elevated risk for autoimmune-related complications with tetracyclines,
6. tetracycline allergy.
7. Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of prolonged minocycline exposure in adult patients with SCD | 12 months (1 year)
  No difference in frequency and/or duration of adverse events between one or both minocycline dose and placebo.

SECONDARY OUTCOMES:
Cognitive Stability | 12 months (1 year)
  Absence of decline and/or improvement in cognitive function measured by NIH Toolbox, for participants on one or both minocycline dose compared to baseline cognitive function and/or to placebo.

IPD SHARING:
Plan to Share IPD: No